CLINICAL TRIAL: NCT02062164
Title: Effectiveness and Safety of Weight Loss Surgery in Adolescents With Extreme Obesity Within a Structured Pre- and Post-surgery Treatment Program, Subproject 3
Brief Title: Weight Loss Surgery in Adolescents With Extreme Obesity
Acronym: YES
Status: Active, not recruiting | Type: Observational
Sponsor: Prof. Dr. Martin Wabitsch (Other)
Collaborators: University of Witten/Herdecke (Other); Charite University, Berlin, Germany (Other); University of Leipzig (Other); Universität Duisburg-Essen (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Martin Wabitsch, Division Chief Pediatric Endocrinology and Diabetology, University of Ulm
Organization: University of Ulm (Other)
Other Study IDs: U1111-1131-4384c; DRKS00004172 (Registry Identifier: Deutsches Register Klinischer Studien); 01GI1120A (Other Grant/Funding Number: German Ministry for Education and Research (BMBF)); U1111-1131-8145 (Other: UTN of overall project)
Record Dates: First submitted 2013-10-22; First posted 2014-02-13 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Extreme Obesity
Keywords: psychosocial, healthcare, co-morbidities, extremely obese adolescents
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of fasting plasma, serum, DNA, urine, visceral and subcutaneous fat will be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- bariatric surgery group: subjects who participate in the overall project and undergo bariatric surgery
  Interventions: Procedure: bariatric surgery
- conservative care group: subjects who participate in the overall project and do not undergo bariatric surgery
  Interventions: Other: conservative care

INTERVENTIONS:
Procedure: bariatric surgery — The intervention takes place in the clinical care setting. The decision for surgery is made by a multidisciplinary team, according to the international guidelines and the recommendations of the German working group on obesity (AGA, www.a.g.a.de). The choice of procedure is made on an individual basis taking into consideration patient inherent factors as well as the recommendations of the operating center. Operations are conducted at certified bariatric centers according to the policies of the German working group on bariatric surgery (CAADIP), and in the context of a structured preparation and follow-up program. The program is offered by a multidisciplinary team (pediatrician, endocrinologist, surgeon, dietician, psychologist/psychiatrist, social worker) and comprises preparation for and education about the surgery and expected lifestyle changes, as well as a structured, multidisciplinary follow-up plan. Subjects sign a contract agreeing to adhere to the recommended follow-up schedule.
  Groups: bariatric surgery group
Other: conservative care — Subjects will be seen by a trained study physician every 6 months. Stuctured health assessments will be conducted, and individual treatment recommendations will be made based on the patients motivation and ability(e.g. inpatient obesity rehab, exercise, dietary or behavioral intervention etc.)
  Groups: conservative care group

SUMMARY:
The use of bariatric surgery in adolescents is controversial. On one side, bariatric surgery is the only effective treatment to achieve sustained weight loss in adults with extreme obesity. Comorbidities are reversed and mortality is reduced. In adolescents, bariatric surgery is equally effective; however, due to the paucity of long-term data, the long-term effects and risks are unknown. Thus, due to surgical risk and ethical implications, bariatric surgery is considered experimental in Germany. Nevertheless, case volumes are increasing.

The aim of this study is to evaluate the benefits and risks of adolescent bariatric surgery in the context of a structured preparation and follow-up program. The study is a subproject of the study "Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care" (DRKS00004172). At 5 German university centers (Ulm, Datteln, Berlin, Essen, Leipzig), youth who undergo bariatric surgery and are participants in the overall project will be enrolled in a structured preparation and follow-up program. The program is designed to improve adherence and compliance and will result in comprehensive follow-up data. In addition to the data gathered in the overall project, subjects participating in subproject 3 will undergo assessments pertinent to bariatric surgery, as proposed in the American Teen-LABS study (http://www.cincinnatichildrens.org/ research/divisions/t/teen-labs/default/). Comparison will be made with BMI matched adolescents who participate in the overall project but do not undergo bariatric surgery.

In November 2014 recruitment for the overall project was completed. However, patients interested in bariatric surgery will still be recruited until September 2016. There assessment will be the same as for patients recruited earlier. However, in an amendment in December 2014, the frequency of assessment via questionnaire was reduced from biannually to annually. In addition, a travel reimbursement of 30€ for each study visit was implemented.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m2 with severe comorbidity or BMI ≥ 40 kg/m2 with relevant comorbidity
* completed longitudinal growth
* stable social surroundings
* exhaustion of conservative treatment
* participation in the project "Adolescents with extreme Obesity"
* adequate compliance and adherence

Exclusion Criteria:

* treatable causative condition
* unstable medical, psychosocial or psychiatric comorbidity
* alcohol or drug abuse
* pregnancy
* contraindication for bariatric surgery

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be recruited from a cohort of young adults and adolescents participating in the "Adolescents with extreme Obesity" Study.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
BMI change from baseline | 1 year postoperative

SECONDARY OUTCOMES:
BMI | every 6 months for 9 years
changes in somatic comorbidity | every 12 months for 9 years
  Will be assessed via standardized physical examination, laboratory and apparative tests, and standardized patient questionnaires.
changes in psychosocial comorbidity | every 12 months for 9 years
  Will be assessed via standardized patient questionnaires.
changes in psychiatric comorbidity | every 12 months for 9 years
  Will be assessed via standardized psychiatric evaluation and standardized and validated patient questionnaires.
peri- und postoperative complications | every 12 months for 9 years
  Will be assessed via physician questionnaires.
vitamin deficiencies | every 6 months for 9 years
  Will be assessed via patient questionnaire and laboratory studies.
adherence with postoperative recommendations on supplements, doctors visits and nutrition | every 12 months for 9 years
  Will be assessed via patient questionnaire.
hunger, food tolerance, gastrointestinal symptoms, dumping | every 12 months for 9 years
  Will be assessed via patient questionnaire.
eating behavior | every 12 months for 9 years
  Will be assessed via validated questionnaire (EDE-Q).
exercise | every 12 months for 9 years
  Will be assessed via validated questionnaire (IPAQ).
changes in quality of life: SF36 | every 12 months for 9 years
  Will be assessed via validated questionnaires (SF36).
changes in quality of life: IWQOL | every 12 months for 9 years
  Will be assessed via validated questionnaires (IWQOL).
schooling, vocation, psychosocial situation, functional impairments | every 12 months for 9 years
  Will be assessed via standardized patient questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wabitsch, Prof. Dr. med., Study Chair — University of Ulm; Susanna Wiegand, Dr. med., Principal Investigator — Charite University, Berlin, Germany; Thomas Reinehr, Prof. Dr. med., Principal Investigator — University of Witten/Herdecke; Johannes Hebebrand, Prof. Dr. med., Principal Investigator — Universität Duisburg-Essen; Wieland Kiess, Prof. Dr. med., Principal Investigator — University of Leipzig; Reinhard Holl, Prof. Dr. med., Principal Investigator — University of Ulm
Locations (5):
- Germany (5):
  - Ambulatory Obesity Program, Charité University, Berlin, Berlin
  - Vestische Kinderklinik, University of Witten/Herdecke, Datteln
  - University Duisburg-Essen, Essen
  - University Hospital Leipzig, Leipzig
  - Dept for Pediatrics and Adolescent Medicine, University of Ulm: Interdisciplinary obesity clinic, Ulm